CLINICAL TRIAL: NCT04212546
Title: Short and Long-Term Effects of Prebiotic, Probiotic and Synbiotic on Appetite and Dietary Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Ankara University (Other)
Responsible Party: Principal Investigator, ZEHRA BUYUKTUNCER, Professor in Nutrition and Dietetics, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: THD-2017-15479
Record Dates: First submitted 2019-12-19; First posted 2019-12-27 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Appetite; Dietary Intake; Body Weight
Keywords: prebiotic; probiotic; synbiotic; hunger and satiety hormones
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Intervention Model Description: This study has two phases. First phase had a randomised, double blind, placebo-controlled crossover study design.
  The second phase had a randomized, double-blind, placebo-controlled parallel study design. The second phase is going to be described below.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control drink (Placebo Comparator): 200 mL milk + 16 g maltodextrin
  Interventions: Other: Control drink
- Test drink (Active Comparator): 200 mL milk + 16 g inulin + Lactobacillus casei [>106 cfu/mL]
  Interventions: Other: Synbiotic test drink

INTERVENTIONS:
Other: Synbiotic test drink — In a healthy male population, participants consumed a synbiotic test drink containing 200 mL milk + 16 g inulin + Lactobacillus casei431 [>106cfu/mL] per day for 21 days with their habitual diet.
  Arms: Test drink
Other: Control drink — In a healthy male population, participants consumed a synbiotic test drink containing 200 mL milk + 16 g maltodextrin per day for 21 days with their habitual diet.
  Arms: Control drink

SUMMARY:
Prebiotics and probiotics are thought to play a role in appetite control and body weight regulation; but little is known about this topic. This study was planned to examine the effects of inulin and Lactobacillus casei 431 on short and long term fasting, satiety, dietary intake, and serum hunger and satiety hormone levels. The study consisted of 2 phases. In the first phase, a double-blind, randomized, crossover study design was used, and it was performed with 16 healthy male participants aged 19-30 years. In this phase, the prebiotic (200mL milk+16g inulin), probiotic (200mL milk + Lactobacillus casei 431 [>106 cfu/mL]+16g maltodextrin), synbiotic (200mL milk+16g inulin + Lactobacillus casei 431 [>106 cfu/mL]) and control (200mL milk+16g maltodextrin) test drinks were consumed with a standard breakfast on four separate test days by one week intervals, and their effects on dietary intake, hunger, satiety and appetite were assessed. The second phase was performed with 21 healthy male participants aged 19-30 years, using a placebo-controlled double-blind, randomized study design. Participants consumed the control (200mL milk+16g maltodextrin) or synbiotic (200mL milk+16g inulin+ Lactobacillus casei [>106 cfu/mL]) test drinks for 21 days with their habitual diet. At the beginning and end of the intervention, blood samples were collected at 0., 30., 60. and 120. minutes following the test day protocol to analyse serum glucose, insulin, ghrelin, obestatin and PYY (peptide tyrosine tyrosine) levels. In addition, dietary intake, hunger, satiety and appetite of participants were compared.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male
* 19-30 years old
* Body mass index (BMI) of 18.5-29.9 kg/m2

Exclusion Criteria:

* Being female
* Being younger than 19 years old or older than 30 years old
* Having a BMI that is lower than 18.5 kg/m2 or higher than 29.9 kg/m2
* Smoking
* Having any metabolic disease
* Losing or gaining weight in the past 3 months
* Following a special diet
* Using any medicine which could affect the outcome of the study
* Having food intolerance and allergies
* Taking regular probiotic or prebiotic foods or supplements
* Not consuming breakfast or lunch regularly
* Being a professional athlete
* Having unhealthy eating attitude that assessed using three factor eating questionnaire (having cognitive restraint score >13, uncontrolled eating score >18, and emotional eating > 6)
* Having depression that was assessed using Beck's Depression Inventory (having a score >9)

Ages: 19 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
Change in dietary energy and nutrient intakes by 3-day dietary record method | At the beginning and end of the intervention (Day 0 and Day 21)
  Energy and nutrients intakes were assessed using a 3-day dietary record method at baseline (including the mean dietary intake of Day -3, Day -2 and Day -1) and at end of the intervention (including the mean dietary intake of Day 19, Day 20 and Day 21).
Change in appetite sensations | 0., 30., 60., 90., 120. and 180. minutes at the beginning and end of the intervention (Day 0 and Day 21)
  Appetite sensation was measured using 100-mm visual analog scale with a minimum value of 0 and a maximum value of 100 at six points including before the breakfast (0.) and following 30., 60., 90., 120. and 180. minutes. Lower scores mean a better outcome.
Change in body weight | At the beginning and end of the intervention (Day 0 and Day 21)
  Body weight was measured

SECONDARY OUTCOMES:
Change in area under the serum glucose concentration versus time curve (AUC) | 0., 30., 60. and 120. minutes at the beginning and end of the intervention (Day 0 and Day 21)
  Serum glucose concentrations were measured at four point including before the breakfast (0.) and following 30., 60. and 120. minutes to provide a curve.
Change in area under the serum insulin concentration versus time curve (AUC) | 0., 30., 60. and 120. minutes at the beginning and end of the intervention (Day 0 and Day 21)
  Serum insulin concentrations were measured at four point including before the breakfast (0.) and following 30., 60. and 120. minutes to provide a curve.
Change in area under the serum obestatin concentration versus time curve (AUC) | 0., 30., 60. and 120. minutes at the beginning and end of the intervention (Day 0 and Day 21)
  Serum obestatin concentrations were measured at four point including before the breakfast (0.) and following 30., 60. and 120. minutes to provide a curve.
Change in area under the serum ghrelin concentration versus time curve (AUC) | 0., 30., 60. and 120. minutes at the beginning and end of the intervention (Day 0 and Day 21)
  Serum ghrelin concentrations were measured at four point including before the breakfast (0.) and following 30., 60. and 120. minutes to provide a curve.
Change in area under the serum PYY concentration versus time curve (AUC) | 0., 30., 60. and 120. minutes at the beginning and end of the intervention (Day 0 and Day 21)
  Serum PYY concentrations were measured at four point including before the breakfast (0.) and following 30., 60. and 120. minutes to provide a curve.
Change in serum fasting adiponectin concentration | At the beginning and end of the intervention (Day 0 and Day 21)
  Serum fasting adiponectin concentrations were measured at the beginning and end of the intervention
Change in dietary energy and nutrient intakes by diet diary method | Day 0, Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11, Day 12, Day 13, Day 14, Day 15, Day 16, Day 17, Day 18, Day 19, Day 20, Day 21
  Energy and nutrients intakes were also assessed using diet diary method during 21-day intervention to confirm the changes assessed by 3-day dietary record.

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Buyuktuncer, PhD, Prof, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Faculty of Health Sciences, Department of Nutrition and Dietetics, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No